CLINICAL TRIAL: NCT04345757
Title: After Cesarean Time Interval for Exercise (ACTIVE) Trial
Acronym: ACTIVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-11021020
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Complications
Keywords: Postpartum wellness; Postoperative activity; Postoperative complication; Postpartum complication
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard instructions (No Intervention): Standard instructions: activity restrictions, including no strenuous exercise, sexual intercourse, or lifting objects greater than 25 pounds for 6 weeks or until evaluation at the 6 week postpartum visit
- Study Group (Experimental): Study group: Structured 10 week exercise protocol
  Interventions: Behavioral: Structured exercise

INTERVENTIONS:
Behavioral: Structured exercise — The exercise program will be designed by a physical therapist (Ms. Patricia Ladis) who specializes in postnatal rehabilitation and will be supervised by sports medicine physicians from the Hospital For Special Surgery (HSS). The structured program will include approximately 10 minutes of core muscle group exercises. They will begin this program 2 weeks after their cesarean section. The study group will perform these exercises 5 times per week.
  Arms: Study Group

SUMMARY:
The purpose of this study is to test whether or not activity restrictions after a cesarean section are warranted and if exercise can improve postpartum wellness. This research study is being done because there is no science-based evidence to support postpartum activity restrictions after cesarean sections.

Participants will be randomly placed into one of the following study groups:

* Standard postpartum and post-operative instructions group: activity restrictions, including no strenuous exercise, sexual intercourse, or lifting objects greater than 25 pounds for 6 weeks or until evaluation at the 6 week postpartum visit
* Study group: Structured 10 week exercise protocol consisting of core strengthening exercises (concentrating on the abdominal, gluteal, and pelvic areas), breathing exercises, and diaphragm exercises.

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman at least 18 years of age
* carrying only one baby at time of delivery
* delivery planned by scheduled cesarean section
* baby of gestational age of > 37 weeks
* no known restrictions to exercise.

Exclusion Criteria:

* woman with pre-existing post operative complications
* medical history with exercise limitations/disabilities
* carrying more than one baby at time of delivery
* delivery (planned by scheduled or emergent) cesarean section with fetal concerns (anomaly, growth restriction, NICU admission, etc)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — all pregnant women
Enrollment: 200 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in wellness | 2, 6, and 10 weeks
  As measured by scores in the completion of the PROMIS GSF assessment.
  The PROMIS GSF assessment uses a method of scoring requiring responses to each item for each participant. Each question usually has five response options ranging in value from one to five. All questions must be answered in order to produce a valid score using the scoring tables. A score of 50 is the average for the United States general population with a standard deviation of 10. A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like Anxiety, a T-score of 60 is one SD worse than average. By comparison, an Anxiety T-score of 40 is one SD better than average. However, for positively-worded concepts like Physical Function-Mobility, a T-score of 60 is one SD better than average while a T-score of 40 is one SD worse than average.

SECONDARY OUTCOMES:
Change in incidence of post operative complications | 2, 6, and 10 weeks
  As measured by number of subjects presenting with any of the following:
  * Wound separation, dehiscence, hernia etc.
  * Re-hospitalization for wound concerns
  * Infection
  * Increased pain, abdominal/core muscle injury
  * Less breastmilk production (adequate-inadequate, Likert scale 1-5)
  * Urinary incontinence
  * Improved fitness
Change in incidence of depression, anxiety, and decreased physical functioning | 2, 6, and 10 weeks
  As measured by scores in the completion of the PROMIS GSF assessment.
  The PROMIS GSF assessment uses a method of scoring requiring responses to each item for each participant. Each question usually has five response options ranging in value from one to five. All questions must be answered in order to produce a valid score using the scoring tables. A score of 50 is the average for the United States general population with a standard deviation of 10. A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like Anxiety, a T-score of 60 is one SD worse than average. By comparison, an Anxiety T-score of 40 is one SD better than average. However, for positively-worded concepts like Physical Function-Mobility, a T-score of 60 is one SD better than average while a T-score of 40 is one SD worse than average.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Kalish, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital Weill Cornell, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No